CLINICAL TRIAL: NCT00351819
Title: Effects of Testosterone Replacement on Pain Sensitivity and Pain Perception in Men With Chronic Pain Syndrome
Brief Title: Effects of Testosterone Replacement on Pain Sensitivity and Pain Perception
Acronym: TAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Shehzad Basaria, ASSOCIATE PROFESSOR, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-27995
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Pain; Hypogonadism
Keywords: Testosterone; Pain; Opioid; Hypogonadism
MeSH Terms: conditions — Pain; Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Androgel (testosterone gel) (Active Comparator): Testosterone replacement therapy
  Interventions: Drug: AndroGel
- Placebo (Placebo Comparator): Placebo gel
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AndroGel — 5g gel, applied once daily to the upper arms, upper back or shoulders.
  Other Names: testosterone gel
  Arms: Androgel (testosterone gel)
Other: Placebo — 5g gel, applied once daily to the upper arms, upper back or shoulders.
  Arms: Placebo

SUMMARY:
Naturally occurring opiates (endorphins) decrease testosterone levels by inhibiting the synthesis of gonadotropin releasing hormone (GnRH) and also inhibiting testosterone synthesis by the testes. Similarly, men with addiction to narcotics and those on exogenous opioids for pain control have decreased serum testosterone levels. Indeed, these men complain of decreased libido, erectile dysfunction and impaired quality of life. Animal studies have shown that gonadectomy results in a decrease in pain threshold in rats and repletion of testosterone elevates that threshold. These observations suggest that testosterone may possess analgesic properties. Hence, the investigators hypothesize that hypogonadism developing in men on opioids results in an increased sensitivity to pain and requirement of higher doses of opioids. In this study, the investigators plan to administer testosterone to men with opioid-induced hypogonadism and evaluate their pain perception, pain sensitivity in response to noxious stimuli and changes in the requirement of opioids in response to testosterone administration.

Hypothesis:

Testosterone replacement in men with opioid-induced hypogonadism will improve pain tolerance, pain perception and quality of life.

Specific aims:

1. To evaluate the effects of testosterone replacement on pain sensitivity, pain tolerance, and pain modulation in men with opioid-induced hypogonadism.
2. To determine the effects of testosterone replacement on health-related quality of life.
3. To determine whether testosterone replacement in hypogonadal men induces changes in the dosage requirements of opioid medications for pain control.

To accomplish our specific aims, the investigators propose a randomized, double blind, placebo-controlled, parallel arm study in which hypogonadal men with non-cancer chronic back pain syndrome on chronic opioids and low testosterone levels (<300 ng/dl) will be randomized to exogenous testosterone replacement therapy vs placebo. Our primary outcome is change in pain tolerance using various external painful stimuli. Secondary outcomes are change in pain sensitivity and modulation, quality of life and opioid requirements.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Age 18 years and older
* Non-cancer chronic pain
* Serum total testosterone level <350 ng/dl
* Consumption of at least 20 mg of hydrocodone (or analgesic equivalent of another opioid) for at least 4 weeks
* Absence of hospitalization in the past 2 months
* No acute illness in the past 2 months
* No current anabolic therapy (growth hormone, DHEA, etc)
* No current use or consumption in the past 2 months of melatonin
* Normal prostate exam
* Normal PSA level

Exclusion Criteria:

* Cancer-related chronic pain
* Liver enzymes > 3 times upper limit of normal
* Serum creatinine > 2 times upper limit of normal
* Neurological disease
* Active psychiatric illness
* Any addictive drug use
* Alcoholism (>3 drinks/day)
* Patients currently receiving melatonin or anabolic agents
* Hospitalization in the past 2 months
* Acute illness in the past 2 months
* Consumption of < 20 mg of hydrocodone (or analgesic equivalent of another opioid)
* Severe BPH
* PSA > 4.0 ng/ml
* Prostate cancer
* Breast cancer

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shehzad Basaria, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhasin S, Travison TG, O'Brien L, MacKrell J, Krishnan V, Ouyang H, Pencina K, Basaria S. Contributors to the substantial variation in on-treatment testosterone levels in men receiving transdermal testosterone gels in randomized trials. Andrology. 2018 Jan;6(1):151-157. doi: 10.1111/andr.12428. Epub 2017 Oct 5. PMID 28981994
- [Derived] Gagliano-Juca T, Icli TB, Pencina KM, Li Z, Tapper J, Huang G, Travison TG, Tsitouras P, Harman SM, Storer TW, Bhasin S, Basaria S. Effects of Testosterone Replacement on Electrocardiographic Parameters in Men: Findings From Two Randomized Trials. J Clin Endocrinol Metab. 2017 May 1;102(5):1478-1485. doi: 10.1210/jc.2016-3669. PMID 27992261
- [Derived] Basaria S, Travison TG, Alford D, Knapp PE, Teeter K, Cahalan C, Eder R, Lakshman K, Bachman E, Mensing G, Martel MO, Le D, Stroh H, Bhasin S, Wasan AD, Edwards RR. Effects of testosterone replacement in men with opioid-induced androgen deficiency: a randomized controlled trial. Pain. 2015 Feb;156(2):280-288. doi: 10.1097/01.j.pain.0000460308.86819.aa. PMID 25599449

RESULTS

PARTICIPANT FLOW:
Groups:
- Androgel (Testosterone Gel): Testosterone replacement therapy
  Androgel (testosterone gel): 5g gel, applied once daily to the upper arms, upper back or shoulders.
Period: Overall Study
Arm/Group | Androgel (Testosterone Gel) | Placebo
Started | 43 | 41
Completed | 36 | 29
Not Completed | 7 | 12
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Elevated PSA | 1 | 1
Not completed — Traumatic ankle fracture | 1 | 0
Not completed — Unprofessional behavior | 1 | 0
Not completed — Non-compliance | 0 | 1
Not completed — Incarcerated | 0 | 1
Not completed — Enrolled in another trial | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Androgel (Testosterone Gel) | Placebo | Total
Number analyzed (Participants) | 36 | 29 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (9) | 50 (6) | 49 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 29 | 65
Region of Enrollment [Number; unit: participants]
  United States | 36 | 29 | 65
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 32.0 (7.0) | 33.4 (8.0) | 32.6 (7.4)
Opioid dose (morphine equivalent) [Mean (Standard Deviation); unit: mg] | 114 (176) | 76 (139) | 97 (161)
Time on opioids [Mean (Standard Deviation); unit: months] | 54 (48) | 40 (54) | 48 (50)
Total testosterone [Mean (Standard Deviation); unit: ng/dL] | 221 (87) | 237 (97) | 228 (91)
Free testosterone [Mean (Standard Deviation); unit: pg/mL] | 44.1 (22.6) | 43.6 (19.3) | 43.9 (21.0)
Sex hormone binding globulin [Mean (Standard Deviation); unit: nmol/L] | 39.3 (31.4) | 37.7 (14.5) | 38.6 (25.2)
Luteinizing hormone [Mean (Standard Deviation); unit: U/L] | 2.8 (1.9) | 3.8 (2.4) | 3.2 (2.2)
TNF-Alpha [Mean (Standard Deviation); unit: pg/mL] | 1.8 (0.6) | 2.2 (2.7) | 2.0 (1.9)
IL-6 [Mean (Standard Deviation); unit: pg/mL] | 2.6 (2.8) | 2.8 (2.9) | 2.7 (2.8)
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 15 [13 to 16] | 14 [13 to 15] | 15 [13 to 15]
Hematocrit [Median (Inter-Quartile Range); unit: %] | 44 [40 to 46] | 43 [39 to 45] | 43 [40 to 45]
Brief Pain Inventory (BPI) questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Brief Pain Inventory (BPI) is a self-administered questionnaire that measuring chronic pain. The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score assesses the severity of pain on a continuous scale from 0 (no pain) to 10 (severe pain). The pain interference score corresponds to the item on pain interference, ranging from 0 (does not interfere) to 10(completely interferes). The total score (ranging from 0-20) is the sum of the pain severity score and pain interference score. Higher scores represents severer and more interfering pain.
  units on a scale
    Total | 11.5 (3.2) | 10.4 (3.1) | 11.0 (3.2)
    Severity | 5.7 (1.5) | 5.5 (1.7) | 5.6 (1.6)
    Interference | 5.8 (2.2) | 4.9 (1.8) | 5.4 (2.1)
Algometer-induced pressure pain [Mean (Standard Deviation); unit: kPa/cm2] — A digital pressure algometer at the trapezius muscle and the metacarpophalangeal joint of the thumb was used to measure pressure pain thresholds. Higher values represent a better tolerance of pressure pain.
  kPa/cm2
    Trapezius | 341 (116) | 353 (197) | 347 (157)
    Thumb | 369 (125) | 383 (185) | 375 (155)
Weighted pinprick stimulator-induced mechanical pain [Mean (Standard Deviation); unit: watt] — Weighted pinprick stimulators are used to assess mechanical pain. Lower values represent better tolerance of pain.
  watt
    First stimulus | 12.0 (13.0) | 8.0 (7.4) | 10.2 (11.0)
    10th stimulus | 27.0 (20.6) | 18.6 (19.5) | 23.2 (20.4)
Ice water-induced cold pain and its after-sensation [Mean (Standard Deviation); unit: seconds] — Cold-pressor tests measure cold-induced pain and its sensation. Time was measured when a participant reached pain tolerance in cold water and after sensation. Higher values of time in Cold pain tolerance and lower values of time in Cold pain after-sensation (30 seconds) represent better tolerance of pain.
  seconds
    Cold pain tolerance | 40.1 (33.4) | 53.3 (51.3) | 46.1 (42.7)
    Cold pain after sensation: 30s | 16.7 (19.2) | 13.8 (18.0) | 15.4 (18.5)
Sexual Function as assessed by International Index of Erectile Function (IIEF) [Mean (Standard Deviation); unit: units on a scale] — IIEF is a validated, 15-item questionnaire that assesses 5 domains of sexual function: erectile function (range 1-30), orgasmic function (range 0-10), sexual desire (range 2-10), intercourse satisfaction (range 0-15), and overall sexual satisfaction (range 2-10). Each question was answered on a 6-point or 5-point scale from 0/1 to 5 (best) with a total possible score (sum of 5 domains) range of 5 to 75 with higher scores representing better function.
  units on a scale
    Total score | 44.6 (19.0) | 41.1 (21.7) | 43.0 (20.2)
    Erectile function | 18.8 (9.2) | 16.8 (10.6) | 17.9 (9.8)
    Orgasmic function | 6.5 (3.5) | 6.1 (3.6) | 6.3 (3.6)
    Sexual desire | 5.5 (2.5) | 6.2 (2.1) | 5.8 (2.3)
    Intercourse satisfaction | 8.2 (4.6) | 7.1 (5.6) | 7.7 (5.1)
    Overall satisfaction | 4.9 (2.5) | 5.0 (2.9) | 4.9 (2.7)
Health Quality of Life (QoL) as assessed by Short Form 36 (SF-36) [Mean (Standard Deviation); unit: units on a scale] — The SF-36 measures 8 domains of the QoL: physical function, bodily pain, vitality, role limitations due to physical problems, general health perceptions, emotional well-being, social function, and role limitations due to emotional problems. Each domain is scored separately from 0 to 100 with higher scores representing better health-related QoL.
  units on a scale
    Physical functioning | 41 (22) | 38 (25) | 39 (23)
    Bodily pain | 56 (15) | 55 (17) | 56 (16)
    Role limitations due to physical health problems | 10 (24) | 18 (31) | 13 (27)
    Role limitations due to emotional problems | 39 (45) | 40 (45) | 39 (44)
    Emotional well-being | 60 (16) | 59 (17) | 60 (16)
    Social functioning | 53 (13) | 54 (15) | 54 (14)
    Energry/fatigue | 37 (18) | 37 (18) | 37 (18)
    General health perceptions | 54 (14) | 51 (14) | 52 (14)
Body composition measured by dual energy x-ray absorptiometry [Mean (Standard Deviation); unit: kg]
  Lean mass | 57.4 (7.8) | 60.1 (6.9) | 58.6 (7.5)
  Fat mass | 27.0 (9.7) | 26.8 (9.5) | 26.9 (9.5)
  Total mass | 84.4 (16.1) | 86.8 (13.8) | 85.5 (15.0)
  Appendicular lean mass | 27.4 (4.0) | 28.6 (4.2) | 27.9 (4.1)
  Appendicular fat mass | 11.7 (4.9) | 11.9 (5.1) | 11.8 (5.0)
  Appendicular total mass | 38.3 (7.8) | 39.4 (7.0) | 38.8 (7.4)
Lipid profile [Mean (Standard Deviation); unit: mmol/L]
  Total cholesterol | 4.6 (1.1) | 5.2 (1.2) | 4.9 (1.2)
  LDL | 2.8 (1.0) | 3.2 (0.9) | 3.0 (1.0)
  HDL | 1.0 (0.3) | 1.1 (0.4) | 1.0 (0.3)
  Triglycerides | 2.0 (1.6) | 2.0 (1.2) | 2.0 (1.4)
HbA1c [Mean (Standard Deviation); unit: percentage of glycossylated hemoglobin] | 5.7 (0.01) | 6.2 (0.02) | 5.9 (0.01)
Glucose levels in OGTT [Mean (Standard Deviation); unit: mmol/L]
  Fasting glucose | 5.2 (0.7) | 5.6 (2.6) | 5.3 (1.8)
  OGTT 1-h glucose | 8.4 (2.9) | 8.0 (2.8) | 8.2 (2.8)
  OGTT 2-h glucose | 6.5 (1.9) | 6.0 (2.0) | 6.3 (1.9)
Insulin levels in OGTT [Mean (Standard Deviation); unit: pmol/L]
  Fasting insulin | 64 (66) | 100 (174) | 80 (126)
  OGTT 1-h insulin | 300 (306) | 416 (325) | 351 (317)
  OGTT 2-h insulin | 246 (242) | 311 (293) | 275 (266)
HOMA IR [Mean (Standard Deviation); unit: HOMA IR score] — Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin. HOMA IR was calculated using the formula: glucose * insulin / 22.5
  HOMA IR score | 2.1 (2.1) | 3.3 (5.8) | 2.6 (4.2)
Adiponectin [Mean (Standard Deviation); unit: ug/mL] — Population: Of the completers, 64 men (36 in the testosterone arm and 28 in the placebo arm) had pre and post-intervention data on Adiponectin outcomes.
  ug/mL
    number analyzed (Participants) | 36 | 28 | 64
    (all) | 4.9 (2.7) | 4.5 (1.7) | 4.7 (2.3)
Leptin [Mean (Standard Deviation); unit: ug/L] — Population: Of the completers, 64 men (36 in the testosterone arm and 28 in the placebo arm) had pre and post-intervention data on Leptin outcomes.
  ug/L
    number analyzed (Participants) | 36 | 28 | 64
    (all) | 16 (12) | 18 (17) | 17 (14)
C-reactive protein [Mean (Standard Deviation); unit: mg/L] — Population: Of the completers, 64 men (36 in the testosterone arm and 28 in the placebo arm) had pre and post-intervention data on C-reactive protein outcomes.
  mg/L
    number analyzed (Participants) | 36 | 28 | 64
    (all) | 3.1 (3.5) | 2.7 (2.3) | 2.9 (3.0)
Pain catastrophizing scale (PCS) [Mean (Standard Deviation); unit: units on a scale] — PCS questionnaire measures self-assessment of pain catastrophizing. This questionnaire consists of 13 items on past painful experiences and rate on 5-point scales ranging from 0 (not at all) to 4 (all the time). The PCS yields three subscale scores assessing rumination (range 0-16), magnification (range 0-12), helplessness (range 0-24), and a composite score (sum of three domains, ranging 0-52). Higher score represents worse painful experiences. Population: Of the completers, 62 men (33 in the testosterone arm and 29 in the placebo arm) had pre and post-intervention data on PCS outcomes.
  units on a scale
    Composite score: number analyzed (Participants) | 33 | 29 | 62
    Composite score | 26 (11) | 27 (11) | 27 (11)
    Rumination score: number analyzed (Participants) | 33 | 29 | 62
    Rumination score | 9.5 (4.0) | 9.6 (3.0) | 9.5 (3.6)
    Magnification score: number analyzed (Participants) | 33 | 29 | 62
    Magnification score | 4.7 (3.2) | 5.1 (2.9) | 4.9 (3.1)
    Helplessness score: number analyzed (Participants) | 33 | 29 | 62
    Helplessness score | 11.5 (5.3) | 11.6 (5.1) | 11.6 (5.2)
Insomnia severity index (ISI) [Mean (Standard Deviation); unit: units on a scale] — ISI is comprised of 7 items assesses a participant's perception of insomnia that specifically address the symptoms and consequences of insomnia, as well as the degree of distress caused by sleep quality. Each item is rated on a 5-point scale from 0 (none) to 4 (very severe). Scores from the questions are summed to assign a total score ranging from 0 to 28, where higher score represents worse insomnia problem. Population: Of the completers, 62 men (33 in the testosterone arm and 29 in the placebo arm) had pre and post-intervention data on ISI outcomes.
  units on a scale
    number analyzed (Participants) | 33 | 29 | 62
    (all) | 11.9 (4.7) | 11.6 (4.4) | 11.8 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI) at Week 14
Description: BPI is a self-administered questionnaire that measuring chronic pain. BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score assesses the severity of pain on a continuous scale from 0 (no pain) to 10 (severe pain). The pain interference score corresponds to the item on pain interference, ranging from 0 (does not interfere) to 10(completely interferes). The total score is the sum of the pain severity score and pain interference score, ranging from 0(no pain) to 20 (severe and completely interfered pain).
Time Frame: Week14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 29
units on a scale
  Total score | 10.2 (3.8) | 9.7 (3.3)
  Severity | 5.3 (1.7) | 5.1 (1.6)
  Interference | 5.0 (2.3) | 4.7 (1.9)

2. Primary Outcome: Algometer-induced Pressure Pain at Week 14
Description: A digital pressure algometer at the trapezius muscle and the metacarpophalangeal joint of the thumb was used to measure pressure pain thresholds. Higher values represent a better tolerance of pressure pain.
Time Frame: Week 14 after intervention
Measure: Mean (Standard Deviation); unit: kPa/cm2
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 29
kPa/cm2
  Trapezius | 379.4 (194.7) | 315.9 (151.6)
  Thumb | 409.7 (167.9) | 326.4 (187.3)

3. Primary Outcome: Weighted Pinprick Stimulator-induced Mechanical Pain at Week 14
Description: Weighted pinprick stimulators are used to assess mechanical pain. Lower values represent better tolerance of pain.
Time Frame: Week 14 after intervention
Measure: Mean (Standard Deviation); unit: watts
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 29
watts
  First Stimulus | 10.9 (8.4) | 11.7 (13.2)
  10th Stimulus | 21.9 (17.4) | 22.2 (23.5)

4. Primary Outcome: Ice Water-induced Cold Pain and Its After-sensation at Week 14
Description: Cold-pressor tests measure cold-induced pain and its sensation. Time was measured when a participant reached pain tolerance in cold water and after sensation. Higher values of time in Cold pain tolerance and lower values of time in Cold pain after-sensation (30 seconds) represent better tolerance of pain.
Time Frame: Week 14 after intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 29
seconds
  Cold pain tolenrance | 54.2 (55.9) | 54.1 (50.9)
  Cold pain after sensation: 30s | 13.1 (18.4) | 13.9 (15.1)

5. Secondary Outcome: Sexual Functioning as Assessed by International Index of Erectile Function (IIEF) at Week 14
Description: IIEF is a validated, 15-item questionnaire that assesses 5 domains of sexual function: erectile function (range 1-30), orgasmic function (range 0-10), sexual desire (range 2-10), intercourse satisfaction (range 0-15), and overall sexual satisfaction (range 2-10). Each question was answered on a 6-point or 5-point scale from 0/1 to 5 (best) with a total possible score (sum of 5 domains) range of 5 to 75 with higher scores representing better function.
Time Frame: Week14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 29
units on a scale
  Total score | 51.3 (17.5) | 47.1 (23.1)
  Erectile function | 21.7 (7.9) | 19.2 (10.8)
  Orgasmic funcion | 7.7 (2.9) | 6.4 (3.4)
  Sexual desire | 6.8 (2.1) | 6.3 (2.6)
  Intercourse satisfaction | 9.1 (5.2) | 9.0 (5.4)
  Overall satisfaction | 6.1 (2.5) | 6.1 (3.1)

6. Secondary Outcome: Health Quality of Life (QoL) as Assessed by Short Form 36 (SF-36) at Week 14
Description: The SF-36 measures 8 domains of the QoL: physical function, bodily pain, vitality, role limitations due to physical problems, general health perceptions, emotional well-being, social function, and role limitations due to emotional problems. Each domain is scored separately from 0 to 100 with higher scores representing better health-related QoL.
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 29
units on a scale
  Physical functioning | 42 (19) | 42 (24)
  Bodily pain | 62 (21) | 61 (17)
  Role limitations due to physical health problems | 23 (35) | 22 (29)
  Role limitations due to emotional problems | 56 (42) | 37 (43)
  Emotional well-being | 64 (16) | 63 (15)
  Social functioning | 57 (14) | 54 (13)
  Energy-fatigue | 44 (17) | 40 (18)
  General health perceptions | 55 (12) | 52 (13)

7. Secondary Outcome: Pain Catastrophizing Scale (PCS) at Week 14
Description: PCS questionnaire measures self-assessment of pain catastrophizing. This questionnaire consists of 13 items on past painful experiences and rate on 5-point scales ranging from 0 (not at all) to 4 (all the time). The PCS yields three subscale scores assessing rumination (range 0-16), magnification (range 0-12), helplessness (range 0-24), and a composite score (sum of three domains, ranging 0-52). Higher score represents worse painful experiences.
Time Frame: Values at week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 33 | 29
units on a scale
  Composite score | 20 (12) | 21 (10)
  Rumination score | 7.1 (4.1) | 7.6 (3.1)
  Magnification score | 3.7 (2.8) | 4.1 (2.4)
  Helplessness score | 9.2 (5.8) | 8.4 (4.7)

8. Other Pre Specified Outcome: Total Testosterone Values at Week 14
Description: Total testosterone was measured in a CDC-certified laboratory using an LC-MS/MS method with a sensitivity of 2 ng/dL.
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 33 | 29
ng/dL | 790 (544) | 328 (185)

9. Other Pre Specified Outcome: Free Testosterone Values at Week 14
Description: Free testosterone was calculated using a law of mass action equation.
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 33 | 29
pg/mL | 189 (152) | 65 (36)

10. Other Pre Specified Outcome: Sex Hormone Binding Globulin (SHBG) at Week 14
Description: Sex hormone binding globulin was measured using immunofluorometric assays, with limits of quantification of 2.5 nmol/L.
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 29
nmol/L | 34.6 (18.2) | 35.0 (14.3)

11. Other Pre Specified Outcome: Luteinizing Hormone Values at Week 14
Description: Luteinizing hormone was measured using immunofluorometric assays, with limits of quantification of 0.05 U/L.
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 29
U/L | 1.6 (2.2) | 3.5 (2.3)

12. Other Pre Specified Outcome: Inflammatory Cytokines at Week 14
Description: The pathophysiology of pain is measured by the proinflammatory cytokines interleukin-6 (IL-6) and tumor necrosis factor alpha (TNF-Alpha).
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 29
pg/mL
  IL-6 | 2.4 (2.1) | 2.6 (2.7)
  TNF-Alpha | 1.9 (1.0) | 2.1 (2.4)

13. Other Pre Specified Outcome: Body Composition at Week 14
Description: Body composition was measured using dual-energy X-ray absorptiometry scan.
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 29
kg
  Lean mass | 57.8 (7.5) | 60.9 (5.9)
  Fat mass | 25.7 (8.7) | 27.9 (9.7)
  Total mass | 83.5 (14.8) | 88.7 (12.8)
  Appendicular lean mass | 27.9 (4.1) | 29.4 (3.7)
  Appendicular fat mass | 11.4 (4.7) | 12.1 (4.7)
  Appendicular total mass | 38.6 (7.9) | 40.8 (6.3)

14. Other Pre Specified Outcome: Lipid Profile at Week 14
Description: Serum total cholesterol, triglycerides and high-density lipoprotein (HDL) cholesterol levels were measured by enzymatic assays and standardized to the CDC using the Lipid Research Clinic protocol. Low-density lipoprotein (LDL) cholesterol was calculated using the Friedewald equation.
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 33 | 27
mmol/L
  Total cholesterol | 4.8 (1.2) | 5.1 (1.1)
  LDL: number analyzed (Participants) | 33 | 26
  LDL | 2.9 (1.0) | 3.1 (1.0)
  HDL | 1.0 (0.4) | 1.1 (0.4)
  Triglycerides | 1.8 (1.0) | 1.9 (1.0)

15. Other Pre Specified Outcome: HbA1c at Week 14
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemogobin
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 28
percentage of glycosylated hemogobin | 5.7 (0.01) | 6.1 (0.01)

16. Other Pre Specified Outcome: Glucose Level in Oral Glucose Tolerance Test (OGTT) at Week 14
Description: All participants underwent 75-g oral glucose tolerance test (OGTT) after a 12-h fast, The plasma glucose level were analyzed at baseline and at 60 and 120 min after glucose loading.
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 33 | 25
mmol/L
  Fasting glucose | 5.2 (1.4) | 5.6 (1.4)
  OGTT 1-h glucose: number analyzed (Participants) | 33 | 24
  OGTT 1-h glucose | 8.0 (3.4) | 8.3 (2.4)
  OGTT 2-h glucose: number analyzed (Participants) | 33 | 24
  OGTT 2-h glucose | 6.7 (3.2) | 6.1 (2.6)

17. Other Pre Specified Outcome: Insulin Level in Oral Glucose Tolerance Test (OGTT) at Week 14
Description: All participants underwent 75-g oral glucose tolerance test (OGTT) after a 12-h fast, The insulin level were analyzed at baseline and at 60 and 120 min after glucose loading.
Time Frame: Values at week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 33 | 25
pmol/L
  Fasting insulin | 70 (88) | 110 (149)
  OGTT 1-h insulin: number analyzed (Participants) | 33 | 24
  OGTT 1-h insulin | 279 (181) | 407 (318)
  OGTT 2-h insulin | 231 (210) | 325 (275)

18. Other Pre Specified Outcome: HOMA IR Score at Week 14
Description: Insulin resistance was calculated using the homeostatic model assessment (HOMA) index: glucose * insulin / 22.5.
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: HOMA IR score
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 33 | 25
HOMA IR score | 2.5 (3.6) | 4.2 (5.9)

19. Other Pre Specified Outcome: Adiponectin at Week 14
Description: Total adiponectin was measured using an RIA kit with an interassay CV of 6.9-9.3% and an intra-assay CV of 1.8-6.2% (Millipore).
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 28
ug/mL | 4.8 (3.0) | 4.7 (2.1)

20. Other Pre Specified Outcome: Leptin at Week 14
Description: Leptin levels were measured using ELISA with an interassay CV of 2.6% to 6.2% and in intra-assay CV of 2.6% to 4.6% (Millipore, Billerica, MA, USA).
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 35 | 28
ug/L | 16 (12) | 21 (21)

21. Other Pre Specified Outcome: C-reactive Protein (CRP) at Week 14
Description: High-sensitivity C-reactive protein (Alpco Diagnostics) was measured using a high-sensitivity sandwich ELISA with an intra-assay CV of 5.6%
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 36 | 28
mg/L | 4.2 (4.4) | 3.4 (3.3)

22. Other Pre Specified Outcome: Insomnia Severity Index (ISI) at Week 14
Description: ISI is comprised of 7 items assesses a participant's perception of insomnia. Each item is rated on a 5-point scale from 0 (none) to 4 (very severe). Scores from the questions are summed to assign a total score ranging from 0 to 28, where higher score represents worse insomnia problem.
Time Frame: Week 14 after intervention
Population: All available data expressed as absolute values at week 14.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Androgel (Testosterone Gel) | Placebo
Number analyzed (Participants) | 33 | 29
units on a scale | 10.8 (5.2) | 11.1 (5.1)

ADVERSE EVENTS:
Arm/Group | Androgel (Testosterone Gel) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/43 | 2/41
Other Adverse Events (participants affected / at risk) | 6/43 | 5/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Androgel (Testosterone Gel) (N=43) | Placebo (N=41)
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Wrist arthrodesis (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Androgel (Testosterone Gel) (N=43) | Placebo (N=41)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Headache (Nervous system disorders) | 2 | 3
Fever (General disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No